CLINICAL TRIAL: NCT02544841
Title: Evaluation of Safer Sex Intervention (SSI)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Policy & Research Group (Other)
Collaborators: Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 5 TP1AH000003-02-00 SSI
Record Dates: First submitted 2015-09-04; First posted 2015-09-09 (Estimated); Last update posted 2016-11-08 (Estimated); Status verified 2016-11

CONDITIONS: Teen Pregnancy Prevention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Safer Sex Intervention (SSI) (Experimental): Safer Sex Intervention (SSI) is the treatment condition. SSI is an in-person, individual-level, clinic-based intervention that aims to reduce risky sexual behaviors among sexually active adolescent females.
  Interventions: Behavioral: Safer Sex Intervention (SSI)
- Female Sexual Health (Active Comparator): Female Sexual Health is the control counterfactual condition. It is an individual-level, information-only sex education program that aims to increase participants' knowledge on various topics related to STIs.
  Interventions: Behavioral: Female Sexual Health

INTERVENTIONS:
Behavioral: Safer Sex Intervention (SSI) — Safer Sex Intervention (SSI) is an in-person, individual-level, clinic-based intervention implemented by a female health educator trained in the intervention. It is intended to be implemented in one initial session lasting 30-50 minutes and three booster sessions lasting 10-30 minutes at one, three, and six month intervals.
  Arms: Safer Sex Intervention (SSI)
Behavioral: Female Sexual Health — Female Sexual Health is a knowledge-based intervention that intends to provide information on how STIs are contracted, the consequences of contracting STIs, and how to prevent them. Female Sexual Health includes the information-only component of the first session of SSI and baseline exposure to a health educator but does not include booster sessions.
  Arms: Female Sexual Health

SUMMARY:
The purpose of the study is to determine the impact of the offer to participate in Safer Sex Intervention (SSI) (treatment) relative to the offer to participate in Female Sexual Health (control) on three self-reported sexual behaviors (condom use, other contraceptive use, and frequency of sex) six months after the end of treatment.

DETAILED DESCRIPTION:
The Policy & Research Group (PRG) will be evaluating the Safer Sex Intervention (SSI). The Safer Sex Intervention is based in Social Cognitive Theory, the Transtheoretical Model of Behavior Change, and motivational interviewing. Coupled with skill-building exercises, the intervention is intended to increase knowledge related to risk and safe-sex behaviors, to increase awareness of risk and need for behavior change, to help build self-efficacy to engage in safe-sex behaviors, and, ultimately, to motivate participants to engage in and maintain safe sex practices. The intervention is meant to be delivered in four, one-on-one sessions over the course of six months. Each session is to be conducted in a private setting by a female health educator trained in motivational interviewing and Safer Sex Intervention. The initial or primary intervention session should take approximately 30 to 50 minutes. Subsequent "booster sessions" delivered 1, 3, and 6 months following the initial session are to take 10 to 30 minutes. Booster sessions are intended to sustain any resulting behavior change. The control (counterfactual) condition, Female Sexual Health, was developed specifically for use in this study; it consists of a 30-minute PowerPoint presentation, intended to be delivered in one face-to-face session that provides information about reproductive anatomy and STIs. After the presentation, participants receive free condoms. This is the only session for the control condition; there are no booster sessions. Though there were some variations in consent requirements across sites, there were no differences in the recruitment process between the treatment and control groups. All eligible individuals who provided the proper consent to participate were randomized and enrolled into the study at the time they attended their first scheduled study session. Data were collected via self-administered questionnaires that were scheduled at baseline and six months post treatment (12 months after baseline). The study took place in New Orleans, Louisiana, at five clinics that served young women between the ages of 14 and 19.

ELIGIBILITY:
Inclusion Criteria:

Between the ages of 14-19 Had engaged in sex with a male in the three months prior to enrollment Provide parental consent (if under age 18) and participant assent to participate in the study.

Exclusion Criteria:

Not have previously participated in any of the following pregnancy/HIV prevention programs:

* 4 Real Health
* Becoming a Responsible Teen (BART)
* Healthy Living
* Staying Mature and Responsible Towards Sex (SMARTS)
* Sisters Informing Healthy Living and Empowering (SIHLE)
* Project AIM
* Making Proud Choices
* Be Proud Be Responsible
* Focus on Your Future

Ages: 14 Years to 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 319 (Actual)
Dates: Start 2012-02; Primary Completion 2015-10 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Two questionnaire items measuring consistency of condom use | 6 months after the end of intervention
  The risk outcome is operationalized as the proportion of times in the past three months a person reports having any type of sex without using a condom. The measure is calculated from the following items on the Outcome Questionnaire administered 6 months after the program ends:
  * In total, how many times have you had any type of sex in the past 3 months?
  * Now, think about the number of times that you had any type of sex in the past 3 months. How many of those times did you use condoms? The resulting variable is a continuous proportion with values that range from 0 to 1, where 0 indicates that a person has not engaged in sex without a condom in the past three months, and 1 indicates that the person has engaged in sex without a condom 100% of the times they had sex in the past three months.

SECONDARY OUTCOMES:
Two questionnaire items measuring consistency of contraceptive use | 6 months after end of intervention
  The risk outcome is operationalized as the proportion of times a person reports having sexual intercourse without using any form of birth control (including condoms). The measure is calculated from the following items:
  * In total, how many times have you had sexual intercourse in the past 3 months?
  * In the past 3 months, how many times have you had sexual intercourse without using any of these methods of birth control (options listed)?
  The measure is calculated by dividing the total number of times a person reported having sexual intercourse without using any contraception by the total number of times she reported having sexual intercourse.
One questionnaire item measuring frequency of sexual activity | 6 months after end of intervention
  The risk outcome is operationalized as the number of times in the past three months a person reports having any type of sex.
  The measure is taken directly from the following item:
  • In total, how many times have you had any type of sex in the past 3 months?
  The variable is continuous, with values ranging from 0 to k, where 0= no sexual activity reported in past 3 months and k = number of times sex reported.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Jenner, PhD, Principal Investigator — The Policy & Research Group